CLINICAL TRIAL: NCT01815892
Title: The Determinants of the Effectiveness of the Use of Furosemide in Patients on Dialysis
Brief Title: The Use of Furosemide in Patients on Dialysis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: MBG1234
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis; Response to Furosemide
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Withdrawal of Furosemide (Active Comparator): The patient's Furosemide will be withdrawn
  Interventions: Drug: Withdrawal of furosemide
- Administration of furosemide (Experimental): The patient will receive furosemide 120 mgms daily
  Interventions: Drug: furosemide administration

INTERVENTIONS:
Drug: Withdrawal of furosemide — The patient (previously on furosemide) will have the furosemide stopped for 2 weeks. The interdialytic weight gain, BP and 24 hour urine volume and sodium excretion will be measured
  Other Names: Lasix
  Arms: Withdrawal of Furosemide
Drug: furosemide administration — The patient will receive 120 mgm furosemide daily for 2 weeks and the interdialytic weight gain, BP and 24 hr urine volume and sodium excretion will be measured.
  Other Names: lasix
  Arms: Administration of furosemide

SUMMARY:
Patients often begin dialysis taking diuretics (stimulate the kidney to excrete salt and water). Once on dialysis, these drugs are often continued. Whether these drugs are still needed, or even effective is often unclear.This study,by evaluating the composition of the patients' urine when off the drug, will predict which patients should benefit from the drug. By comparing their 24 hour volume both off and on the drug, the impact of the drug will be established. The results will allow the prediction of which patients, in the future, should take the drug. The hypothesis is: Among dialysis recipients, evaluation of the random urine sodium concentration will help predict the likelihood of a positive response to Furosemide, as manifested by an increased urine volume and sodium excretion.

DETAILED DESCRIPTION:
Patients often begin dialysis on a significant dose of diuretic due to the retention of sodium and water in the predialysis phase of their chronic kidney disease (CKD). The quandary often faced by the care team is whether or not the diuretic should be continued on dialysis, particularly after they have been on dialysis for a period of time. For the appropriate dialysis patient, a daily dose of furosemide,, minimizes the interdialytic weight gain, may result in better blood pressure (BP) control and may lower the risk of heart failure. Furthermore, there may be a favourable impact on cardiac remodeling and cardiac morbidity and mortality. The diuretic may also increase the excretion of potassium, thereby reducing the likelihood of hyperkalemia.

Patients with significant renal sodium reabsorption would be the ones who would be expected to respond to furosemide. Thus patients whose urine [Na] is less than 80 mM are reabsorbing significant amounts of filtered Na (glomerular filtrate [Na] would be between 130 and 140mM) and thus might be expected to respond to furosemide. (This is premised on the assumption that the urine [Na] does not vary much during the day in chronic dialysis recipients, but this will be established during the course of the study.)

The patients Dry Weight will be optimized prior to entry into study according to usual care: this involves integrating BP data, the central venous pressure as assessed by the internal jugular vein, and patient symptoms (eg,dyspnea during the interdialytic interval,prolonged lightheadedness/presyncope/fatigue after dialysis)..

Patients on dialysis who are taking furosemide will be asked to stop their furosemide for 2 weeks, and their dry weight maintained with ultrafiltration on dialysis alone.

After 2 weeks, to establish whether there is any diurnal variation in the urine [Na] they will collect their urine in separate containers, appropriately labeled with the date and time, during the 24 hr period ending pre dialysis after the long interdialytic interval. These collections will also determine whether there is any diurnal variation in [Na], the individual urine [Na], as well as indicate the 24 hour urine volume and Na excretion off the furosemide.

All urine samples will be assayed for the concentration of Na, K, and creatinine, as well as their volume.

Thereafter, each patient will be given furosemide 120 mgm every morning for 2 weeks and they will collect the urine voided with each voiding (labeling with the time voided) in separate containers during the 24 hr period ending pre dialysis after the long interdialytic interval after 2 weeks . These collections will answer whether there is any diurnal variation in [Na] while on furosemide, as well as determine the 24 hour urine volume and Na excretion on the furosemide.

The results will determine whether those patients taking furosemide are indeed benefitting from it (Na, K and H2O excretion) and will help one to predict whether patients not taking furosemide, might indeed benefit from taking it.

At the conclusion of the 2-week period of furosemide therapy, the patient's primary nephrologist will determine the need for continuing this agent and if a decision is made to continue furosemide, the dose would be at the discretion of the nephrologist.

The primary outcome is the increase in urine volume and 24 hour sodium excretion in response to the furosemide therapy

ELIGIBILITY:
Inclusion Criteria:all patients taking Furosemide -

Exclusion Criteria:Patients not willing to give consent

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
24 hour urine sodium and water excretion | 2 weeks
  The patients 24 hour sodium and water excretion on and off the medication (which they had already been taking) will be compared for effectiveness of the drug. The hypothesis is that the urine sodium concentration off the drug, will predict the response and thus be of diagnostic value for other patients

SECONDARY OUTCOMES:
Interdialytic weight gain | 2 weeks
  The interdialytic weight gain on and off the drug will be compared

OTHER OUTCOMES:
The patients' BP on and off the drug will be compared | 2 weeks
  The patients pre dialysis BP as well as the 48 hr ambulatory BP (if the patient is willing) will be compared in both phases of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Marc B Goldstein, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada